CLINICAL TRIAL: NCT01377597
Title: A 3-month, Phase III, Open-label, Single Arm, Multicenter Study Assessing the Efficacy and Safety of 0.5 mg Ranibizumab Monthly Intravitreal Injections as Monotherapy in Patients With Visual Impairment Due to Macular Edema Secondary to Branch or Central Retinal Vein Occlusion (RVO)
Brief Title: Efficacy and Safety of Ranibizumab in Japanese Patients With Retinal Vein Occlusion
Acronym: RVO in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002E2301
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Retinal Vein Occlusion
Keywords: retinal vein occlusion; branch retinal vein occlusion; central retinal vein occlusion; visual impairment; macular edema; ranibizumab
MeSH Terms: conditions — Retinal Vein Occlusion; Vision Disorders; Macular Edema | interventions — Ranibizumab

ARMS (1):
- ranibizumab intravitreal injection (Experimental)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab

SUMMARY:
The purpose of this study is to provide efficacy and safety data of 3 consecutive monthly intravitreal injections with 0.5 mg ranibizumab in Japanese patients with visual impairment due to macular edema secondary to retinal vein occlusion (BRVO or CRVO) to support the applicability of the phase III study results of BRAVO and CRUISE in this indication, in the Japanese ethnic patients.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients diagnosed with visual impairment exclusively due to macular edema secondary to either branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO) Diagnosis within 12 months prior to Visit 1
* Best-corrected visual acuity (BCVA):
* CRVO: BCVA score ≥24 and ≤73 letters ETDRS (approx. Snellen equivalent of 20/320 and 20/40) at Visit 1 and 2
* BRVO: BCVA score ≥19 and ≤73 letters ETDRS (approx. Snellen equivalent of 20/400 and 20/40) at Visit 1 and 2

Exclusion Criteria:

* Pregnant or nursing women
* History of stroke
* Uncontrolled blood pressure
* Active ocular infection or intraocular inflammation in either eye
* Uncontrolled glaucoma in either eye
* Neovascularization of the iris or neovascular glaucoma in either eye
* Prior episode of RVO more than 12 months prior to Visit 1 in the study eye
* Use of any systemic anti-VEGF drugs within 6 months prior to Visit 2
* Prior treatment with any anti-angiogenic drugs within 3 months prior to Visit 2 in either eye
* Prior panretinal laser photocoagulation within 3 months prior to Visit 2 in the study eye
* Prior focal/grid laser photocoagulation within 4 months prior to Visit 2 in the study eye
* Use of intra-/peri-ocular corticosteroids within 3 months prior to Visit 1 in the study eye
* Use of any intra-ocular corticosteroid implants in the study eye

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measure: Efficacy of 3 consecutive monthly intravitreal injections with 0.5 mg ranibizumab as assessed by the mean average change in best-corrected visual acuity (BCVA) from Month 1 through Month 3 compared to baseline | 3 months

SECONDARY OUTCOMES:
Measure: Efficacy of monthly ranibizumab injections as assessed by the mean BCVA change from baseline over time to Month 3, by visit | 3 months
Measure: Efficacy of monthly ranibizumab injections as assessed by the mean change in central subfield thickness (CSFT) of the retina from baseline over time to Month 3 | 3 months
Measure: Efficacy of monthly ranibizumab injections as assessed by the proportion of patients achieving BCVA improvement of ≥1, ≥5, ≥10, ≥15, and ≥30 letters from baseline to Month 3 | 3 months
Measure: Efficacy of monthly ranibizumab injections as assessed by the proportion of patients with a BCVA loss of <15 letters from baseline to Month 3 | 3 months
Measure: Safety of monthly ranibizumab injections as assessed by the type, frequency and severity of adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharma AG, Study Director — Novartis Pharmaceuticals
Locations (7):
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Ohtsu, Shiga

REFERENCES:
- [Result] Kamei M, Terasaki H, Yoshimura N, Shiraga F, Ogura Y, Grotzfeld AS, Pilz S, Ishibashi T. Short-term efficacy and safety of ranibizumab for macular oedema secondary to retinal vein occlusion in Japanese patients. Acta Ophthalmol. 2017 Feb;95(1):e29-e35. doi: 10.1111/aos.13196. Epub 2016 Sep 22. PMID 27654837